CLINICAL TRIAL: NCT00875953
Title: Harmonic Scalpel vs. Electrocautery in Modified Radical Neck Dissection: A Single Blinded Prospective Randomized Trial
Brief Title: Use of the Harmonic Scalpel in Neck Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Joseph C. Dort BSc, MSc, MD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCENT003
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2009-04

CONDITIONS: Neck Dissection
Keywords: squamous cell carcinoma; head and neck cancer; neck dissection
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dissection (Active Comparator): standard neck dissection technique: scalpel and cautery.
  Interventions: Procedure: standard neck dissection
- Harmonic Scalpel (Experimental): Harmonic scalpel used in neck dissection.
  Interventions: Procedure: Harmonic Scalpel Dissection

INTERVENTIONS:
Procedure: standard neck dissection — standard surgical technique
  Arms: Standard dissection
Procedure: Harmonic Scalpel Dissection — harmonic scalpel used for neck dissection after flaps are raised.
  Other Names: ethicon harmonic scalpel used
  Arms: Harmonic Scalpel

SUMMARY:
Neck dissection is the main technique used by head and neck surgeons to treat known or suspected metastatic cancer to the neck. The traditional radical neck dissection was effective at treating metastatic cancer to the neck however the downside to this technique was significant morbidity. Since the early 1960's there has been several proposed techniques to treat metastatic head and neck cancer that involves preserving important anatomical structures in the neck. The disadvantage to these techniques are that they require meticulous dissection and can lead to bleeding and an increase in operative time. One particular tool that has been proposed in other surgical subspecialties, including head and neck surgery, is the harmonic scalpel. Using this tool, tissue dissection and vessel occlusion at the same time can occur with a reduced thermal damage to the surrounding tissue when compared to traditional cautery. In this study, our purpose is to determine if the harmonic scalpel will lead to a decrease in blood loss and operative time in patients undergoing a modified radical neck dissection compared to electrocautery.

Hypothesis: Use of the harmonic scalpel as a surgical adjunct will reduce operative time for neck dissection and will reduce intraoperative blood loss.

DETAILED DESCRIPTION:
Patients who are referred to either the clinic of Dr. Joseph Dort or Dr. Wayne Matthews and are deemed to benefit from a modified radical neck dissection alone or as part of treatment for head and neck cancer will be given an opportunity to be a subject in this study. Once informed consent for both the surgery and the study is obtained, the lead author will be contacted and randomization will occur using a computer generated block-randomization allocation. The neck dissection will be carried out in the operating room using either electrocautery (control group) or harmonic scalpel (experimental group). The primary outcomes, blood loss (mLs) and operative time (minutes) will be assessed at the time of surgery. The blood loss in milliliters will be calculated using suction canister output, weight of sponges and irrigation used. The operative time in minutes will be calculated between the beginning of the actual neck dissection to the completion of the neck dissection defined as the removal of the surgical specimen and hemostasis of the surgical field. Intraoperative complications, namely vascular, nerve damage and lymphatic damage will be assessed at the time of surgery. Post-operative complications, both early and late will be assessed after the surgery using the Clavien post-operative complication scale. In addition, the length of time that operative drains are left in the neck will be measured with all drains being removed when their 24 hour drain output is less than 20 mls. Patients will then be followed up 2 weeks after their hospital discharge in the surgeon's clinic or the Tom Baker Cancer Centre.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* undergoing neck dissection (levels I-IV)

Exclusion Criteria:

* no prior head and neck surgery
* no prior head and neck cancer
* no prior head and neck radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
operative blood loss | intraoperative
Operating Time | at end of the procedure

SECONDARY OUTCOMES:
wound drainage | 48 hours
wound infection | 48 hours, 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Dort, BSc, MSc, MD, Principal Investigator — University of Calgary - Faculty of Medicine
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada